CLINICAL TRIAL: NCT01102803
Title: Evaluation of the Effects of Post-Session Administration of D-cycloserine On Exposure Therapy Outcomes
Brief Title: D-Cycloserine to Enhance Cognitive Behavioral Therapy (CBT) for Acrophobia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Principal Investigator, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS09-81
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2012-12

CONDITIONS: Phobic Disorders
Keywords: Phobias; Anxiety Disorders; D-Cycloserine; Phobic Disorders; Mental Disorders; Heights; Acrophobia
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders; Mental Disorders; Acrophobia | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Participants will receive placebo augmented cognitive behavioral therapy
  Interventions: Behavioral: Individual Cognitive Behavioral Therapy (CBT); Drug: Placebo
- D-Cycloserine (Experimental): Participants will receive D-Cycloserine augmented cognitive behavioral therapy
  Interventions: Behavioral: Individual Cognitive Behavioral Therapy (CBT); Drug: D-Cycloserine

INTERVENTIONS:
Behavioral: Individual Cognitive Behavioral Therapy (CBT) — The aim of CBT is to help participants become more comfortable with heights situations. Participants will receive 2 sessions over two weeks of individual CBT.
  Other Names: CBT; DCS
Drug: D-Cycloserine — D-Cycloserine
  Arms: D-Cycloserine
Drug: Placebo — Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to investigate the utility of post-session administration of D-cycloserine to enhance fear extinction in a sample of people with acrophobia who will be treated with CBT.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18-65 years of age with a psychiatric diagnosis of acrophobia defined by DSM-IV criteria.
2. Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

1. A lifetime history of bipolar disorder, schizophrenia, psychosis, delusional disorders or obsessive-compulsive disorder; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance (amphetamines, benzodiazepines, barbiturates, cocaine metabolites, marijuana, narcotics, and sedative hypnotics) abuse or dependence or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
2. Patients with posttraumatic stress disorder and panic disorder within the past 6 months are excluded. Entry of patients with other mood or anxiety disorders will be permitted in order to increase accrual of a clinically relevant sample. Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Patients must be off concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) for at least 2 weeks prior to initiation of randomized treatment.
4. Significant personality dysfunction likely to interfere with study participation.
5. Serious medical illness or instability for which hospitalization may be likely within the next year.
6. Patients with a current or past history of seizures.
7. Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
8. Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration directed specifically toward treatment of acrophobia is excluded. Prohibited psychotherapy includes CBT therapy focusing on exploring specific, dynamic causes of the phobic symptomatology and provides management skills. General supportive therapy initiated > 3 months prior is acceptable.
9. Prior non-response to adequately delivered exposure (i.e., as defined by the patient's report of receiving specific and regular exposure assignments as part of a previous treatment) will exclude participants from the study.
10. Patients with a history of head trauma causing loss of consciousness, seizure or ongoing cognitive impairment.
11. Patients receiving isoniazid.
12. Patients unable to understand study procedures and participate in the informed consent process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, Ph.D., Principal Investigator — Southern Methodist University
Locations (1):
- Southern Methodist University, Dallas, Texas, United States

REFERENCES:
- [Derived] Smits JA, Rosenfield D, Otto MW, Powers MB, Hofmann SG, Telch MJ, Pollack MH, Tart CD. D-cycloserine enhancement of fear extinction is specific to successful exposure sessions: evidence from the treatment of height phobia. Biol Psychiatry. 2013 Jun 1;73(11):1054-8. doi: 10.1016/j.biopsych.2012.12.009. Epub 2013 Jan 16. PMID 23332511
- [Derived] Tart CD, Handelsman PR, Deboer LB, Rosenfield D, Pollack MH, Hofmann SG, Powers MB, Otto MW, Smits JA. Augmentation of exposure therapy with post-session administration of D-cycloserine. J Psychiatr Res. 2013 Feb;47(2):168-74. doi: 10.1016/j.jpsychires.2012.09.024. Epub 2012 Oct 23. PMID 23098672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (N = 29; Mean age = 33.38) with acrophobia were recruited from Southern Methodist University and the greater Dallas area from 2009 to 2011.
Pre-assignment Details: 76 individuals were assessed for eligibility, of which 47 were excluded due to not having a diagnosis of acrophobia (n=37) or declining participation (n=10). 29 individuals were randomized and no participants were excluded after enrollment but prior to group assignment.
Groups:
- Sugar Pill: Participants will receive sugar pill placebo augmented cognitive behavioral therapy
- D-Cycloserine: Participants will receive D-Cycloserine (50mg) augmented cognitive behavioral therapy
Period: Baseline to Post-Treatment
Arm/Group | Sugar Pill | D-Cycloserine
Started | 14 | 15
Completed | 11 | 15
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0
Period: Post to Follow-Up
Arm/Group | Sugar Pill | D-Cycloserine
Started | 11 | 15
Completed | 10 | 12
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | D-Cycloserine | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.71 (16.81) | 29.33 (14.67) | 33.8 (15.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Acrophobia Questionnaire With Avoidance (AAVQ)
Description: Self-report measure that assesses fear and avoidance of a variety of heights situations. This questionnaire (Cohen, 1977) describes 20 situations and assesses levels of avoidance (0-3) and anxiety (0-6). These scales widely used measure of acrophobia with adequate retest reliability (r = .82-.86) and validity (Baker et al., 1973). Higher scores indicate higher levels of avoidance/anxiety (i.e., worse outcome). All subscales are summed for a total score. AAVQ will be assessed at each visit throughout the 2 month protocol. The minimum score is 0, the maximum is 90.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DCS+CBT Treatment: Participants receiving DCS augmented CBT
- Placebo+CBT Treatment: Participants receiving PL augmented CBT
Arm/Group | DCS+CBT Treatment | Placebo+CBT Treatment
Number analyzed (Participants) | 15 | 14
units on a scale | 9.00 (7.41) | 12.38 (9.72)

2. Secondary Outcome: Attitudes Towards Heights Questionnaire (ATHQ)
Description: Self-report measures that assesses thoughts and feelings towards heights situations. This questionnaire (Abelson and Curtis, 1989) includes six heights situations and assesses attitudes toward these situations using a 0-10 scale. Higher scores indicate a worse outcome and total scores are summed over subscales. Will be assessed at each visit throughout the 2 month protocol. The minimum score is a 0; the maximum is a 60.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | D-Cycloserine
Number analyzed (Participants) | 15 | 14
units on a scale | 45.67 (8.53) | 47.71 (12.98)

3. Secondary Outcome: Clinical Global Improvement Scale (CGI)
Description: Clinician-rated measure of improvement in acrophobia symptoms and severity. Will be assessed at each visit throughout the 2 month protocol. The CGI-S and CGI-I are widely used measures of global psychopathology severity and improvement initially developed for the study of psychotropic drugs (Guy, 1970). In order to obtain CGI ratings, the therapists (blind to study condition) interviewed the participant and used the SCID (including the specific phobia module) as well as the additional measures of acrophobia symptoms (BAT, AAQ, AAVQ, and ATHQ). In the current study, response was defined as either "very much improved" or "much improved" on CGI-I (score ≤ 2). Remission was defined as either "normal" or "minimally ill" on CGI-S (score ≤ 2). The minimum rating is a 1 and the highest is a 7. Lower scores indicate a better outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | D-Cycloserine
Number analyzed (Participants) | 15 | 14
units on a scale | 2.27 (.96) | 2.00 (.89)

4. Secondary Outcome: Behavioral Avoidance Test (BAT)
Description: During the initial screen, at post-treatment, and at follow-up, participants underwent a behavioral avoidance test in the virtual reality height environment. Participants reported on a 0-100 scale (100 being the most intense fear) their SUDS for floors 1, 2, 3, 4, 9, 19 of the virtual glass elevator and balconies. This test has been used successfully as a measure of treatment gains in previous studies of acrophobia research (Ressler et al., 2004). For the outcome analyses, we included the level of fear reported at the highest floor of the virtual elevator environment (19th floor). Higher scores indicate a worse outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | D-Cycloserine
Number analyzed (Participants) | 15 | 14
units on a scale | 29.73 (25.67) | 35.55 (25.18)

ADVERSE EVENTS:
Groups:
- DCS+CBT: CBT augmented with DCS (50mg)
- Pill Placebo + CBT: CBT augmented with sugar pill placebo
Arm/Group | DCS+CBT | Pill Placebo + CBT
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
Sample may not have been severe enough to see an effect of DCS; there may have been a ceiling effect; there was no pre-session pill administration; assessors were blind but not independent; only one dose of DCS was examined

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No